CLINICAL TRIAL: NCT07300488
Title: Randomized, Controlled, Open-Label, Multicenter Phase Ⅱ/Ⅲ Seamless Adaptive Design Registration Clinical Trial of Pracytarabine Versus Regorafenib for Advanced Hepatocellular Carcinoma After Failure of Targeted Drugs and Immune Checkpoint Inhibitors or Dual Immune Checkpoint Inhibitors Therapy
Brief Title: Efficacy and Safety of Pracytarabine Versus Regorafenib in the Treatment of Patients With Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB07133-2025-01
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: HCC
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pracytarabine (Experimental): Treatment with 1200 mg/m²/d Pracytarabine
  Interventions: Drug: Pracytarabine
- regorafenib (Active Comparator): Treatment with regorafenib 160 mg once daily
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: Pracytarabine — Pracytarabine 1200 mg/m²/d, administered as a continuous intravenous infusion for 7 days (Days 1 to 7), followed by a 21-day treatment-free observation period; each treatment cycle is 4 weeks.
  Arms: Pracytarabine
Drug: regorafenib — Regorafenib 160 mg, once daily, administered continuously for 3 weeks followed by 1 week of rest, i.e., each cycle is 4 weeks.
  Arms: regorafenib

SUMMARY:
This is a Phase 2/3 study evaluating the efficacy and safety of Pracytarabine versus regorafenib in patients with advanced hepatocellular carcinoma (HCC) who have experienced treatment failure with standard systemic therapies involving targeted drugs and immune checkpoint inhibitors, or dual immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, regardless of gender.
2. Diagnosed with HCC either by histopathological and/or cytological examination meeting pathological diagnostic criteria, or in line with the clinical diagnostic criteria of the aforementioned guidelines.
3. Unresectable or metastatic HCC, and have experienced treatment failure with targeted drugs and immune checkpoint inhibitors.
4. Child-Pugh liver function score: Class A/B (≤7 points).
5. Expected survival time ≥ 3 months.
6. ECOG performance status 0 or 1.
7. Barcelona Clinic Liver Cancer (BCLC) stage B or C.
8. No severe involvement of the portal vein, and no invasion of the hepatic vein, superior vena cava, or inferior vena cava.

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
2. Previous history of liver or other organ transplantation.
3. Has participated in another clinical study within 4 weeks prior to the first dose.
4. Has a known history of, or any evidence of CNS metastases.
5. Clinically symptomatic or recurrently drained pleural effusion, pericardial effusion, or ascites.
6. History of bleeding event due to esophageal and/or gastric varices within 3 months prior to the first dose of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
9-month Overall Survival (OS) rate | Up to 12 months
  9-month Overall Survival (OS) rate：The proportion of the total number of subjects who survived for 9 months from randomization.

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed by investigator per RECIST v1.1 | Up to 12 months
  PFS is defined as the time from randomization till the first documented disease progression (Per RECIST v1.1 assessed by the investigator) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Tianyinshan Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No